CLINICAL TRIAL: NCT06105541
Title: At-Home Transcutaneous Auricular Neuromodulation for Hypermobile Ehlers Danlos Syndrome
Brief Title: Hypermobile Ehlers-Danlos Syndrome - Transcutaneous Auricular Neuromodulation
Acronym: hEDS-tAN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Jeffrey Borckardt, Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00128818
Record Dates: First submitted 2023-08-09; First posted 2023-10-27 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Hypermobile Ehlers-Danlos Syndrome; Hypermobile Spectrum Disorder; Ehlers-Danlos Syndrome
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3; Ehlers-Danlos Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two paralell groups:
  Group 1: Double-blind phase Active, Open-label phase Active Group 2: Double-blind phase Sham, Open-label phase Active
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 2 Weeks Sham tAN followed by 2 Weeks Active tAN (Experimental): Participants will be randomized to receive 2 weeks of at-home, self-administered sham Transcutaneous Auricular Neurostimulation (tAN), followed by 2 weeks of at-home, self-administered active Transcutaneous Auricular Neurostimulation (tAN).
  Interventions: Device: Transcutaneous Auricular Neurostimulation
- Four Weeks of Active Transcutaneous Auricular Neurostimulation (Experimental): Participants will be randomized to receive 2 weeks of at-home, self-administered active Transcutaneous Auricular Neurostimulation (tAN), followed by 2 additional weeks of at-home, self-administered active Transcutaneous Auricular Neurostimulation (tAN)
  Interventions: Device: Transcutaneous Auricular Neurostimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Neurostimulation — Transcutaneous Auricular Neurostimulation (tAN) is a wearable, electrical stimulation device that delivers electricity to specific parts of the human ear.

SUMMARY:
Investigate whether at-home transcutaneous auricular VNS (tAN: transcutaneous auricular neurostimulation) improves a battery of nine key physical and psychological symptoms of a group of hEDS (Hypermobile Ehlers-Danlos Syndrome & Hypermobile Spectrum Disorder) patients (n=30) using a randomized, double blind, sham controlled design. The study team will collect clinical measures at baseline, after a two-week double-blind intervention phase, after a following two-week open-label phase and finally at three months post intervention. The study team will test patients in the following domains: pain, fatigue, sleep, anxiety, depression, quality of life, GI function, immune function and autonomic function.

DETAILED DESCRIPTION:
The intervention we are studying is called transcutaneous auricular neurostimulation (tAN). tAN is simply electrical nerve stimulation administered at the ear which targets both the auricular branch of the vagus nerve (ABVN) and the auricular branch of the trigeminal nerve (ATN). tAN will be administered using a the Spark Sparrow Ascent System that PI Dr. Badran has used in a prior MUSC IRB-Approved Neonatal study and has also been approved for human research applications as a non-significant risk investigational device. The Sparrow Ascent tAN device, as of June 21, 2023, has received FDA 510(k) clearance (K230796) and is indicated as a transcutaneous nerve field stimulator that is intended to be used in both the inpatient and outpatient setting for patients experiencing opioid withdrawal. However in this paradigm we will be using the device as an research device in individuals with EDS, with identical stimulation guidelines that are prescribed and used in the FDA indicated manner.

The Sparrow Ascent tAN System is intended to stimulate branches of the vagus and trigeminal nerves on and/or around the ear. This is based on the first FDA-cleared device that non-invasively stimulates both the vagus and trigeminal nerves. tAN has been shown in multiple clinical trials to reduce pain associated with opioid withdrawal in adults and neonates. The Sparrow Ascent System utilizes a flexible earpiece with embedded hydrogel electrodes that adhere to the skin, the earpiece is disposable after use, and delivers a non-opioid and non-pharmacological therapy. The system is capable of fully customizing stimulation parameters to match each participants' therapeutic requirements. Stimulation parameters on the Patient Controller can be using the interface on the Patient Controller. The Patient Controller delivers electrical stimulation to the earpiece via a removable cable. Patients can modulate therapy intensity by pressing up/down buttons and check therapy status with LED lights. The Sparrow earpiece is applied for each patient to position the electrodes to stimulate three key dermatome regions. These regions are adjacent to several cranial nerves (V, VII, IX, X) and occipital nerves. In particular, the electrodes are located on the cymba concha, on the temporomandibular join region, just anterior to the tragus, and behind the auricle.

In this study, participants will be randomized to receive twice daily (1hr per session) either active- or sham tAN treatment outlined below.

All participants will be randomized to receive either active or sham tAN in the first blinded phase of this trial (2 weeks). Afterwards, all participants, regardless of stimulation condition, will receive 2 additional weeks of active tAN in an open-label arm. Thus participants may receive one of the following:

* 2 weeks active tAN followed by an additional 2 weeks of active tAN
* 2 weeks sham tAN followed by an additional 2 weeks of active tAN

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet the 2017 diagnostic criteria for hEDS or HSD4-5 with persistent symptoms in at least two of the domains to be followed during the intervention (pain, fatigue, sleep, anxiety, depression, quality of life, GI function, autonomic function and immune function)
* Mentally capable of reading, writing, giving consent, and following instructions

Exclusion Criteria:

* MRI-contraindicated implanted medical devices;
* pregnant
* history of seizures
* prior history of trauma or damage to ear

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2026-02-04 (Estimated)

PRIMARY OUTCOMES:
Ehlers-Danlos Syndrome Symptom Battery | 16 weeks
  The investigators have created an Ehlers-Danlos Syndrome Symptom Battery that measures a variety of different primary and secondary symptoms associated with Ehlers-Danlos Syndrome, including: Pain, Fatigue, Sleep, Anxiety, Depression, Quality of Life, and Gastrointestinal issues

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States